CLINICAL TRIAL: NCT06749938
Title: A Holistic Intervention Approach to Maximize Quality of Life for Cancer Survivors
Brief Title: Holistic Intervention for Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Daniel Hughes, Assistant Professor, The University of Texas Health Science Center at San Antonio
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC2019-0637H
Record Dates: First submitted 2024-12-11; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Cancer
Keywords: yoga; cancer survivorship; functionality; quality of life; aging; mobility
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Holistic Intervention (Experimental): The holistic intervention comprises of Aerobic Exercise Prescription, Yoga and Meditation Exercise, Diet Intervention, and Psychosocial Support
  Interventions: Other: Holistic Intervention

INTERVENTIONS:
Other: Holistic Intervention — * Aerobic Exercise Prescription. Each participant will be given instruction on an exercise program to progress to perform a total of 150 minutes/wk of moderate-vigorous aerobic activity (including any yoga practice they choose to do) with two days of strengthening exercises using exercise bands.
  * Yoga Protocol and Meditation Exercise. Participants will be asked to practice three 75-min session days per week. The program will focus on developing breath and body awareness/control (pranayama), focused concentration, meditation, muscular strength, muscular endurance, and mobility (flexibility) training that involves the mind body spirit connection.
  * Diet Intervention. Coaching for diet modification will be incorporated into the psychosocial support messaging.
  * Psychosocial Support. Motivational strategies to enhance exercise compliance comprise of electronic messaging using the BlueJay Mobile-Health, (Livermore, CA). This tele-health HIPPA compliant allows private communication.
  Other Names: holistic approach

SUMMARY:
There are many components to defining a cancer survivor's true quality of life. Quality of life (QOL) can be conceptualized as the maximum realization of an individual's potential outcomes of the physical, mental and spiritual aspects defining a human being. These levels of optimization are often limited within certain bounds by a survivor's medical history such as the cancer experience; functional capacities; dietary choices, connectedness and cognitive processing, e.g. perceptions about life situations such as stressors. Often, in intervention studies and within traditional Western medicine practice, focus on optimizing outcomes for cancer survivors is often "siloed", overly focusing on only one aspect of QOL and not accounting for improving other equally important aspects of QOL. A holistic approach, tailored to the unique aspects for that particular survivor, is needed to maximize the individuals overall QOL. Precision scientific data needs to be collected, as well as the cancer survivor's self-report perceptions (qualitative) to truly understand the individual's level of QOL. Thus, both quantitative and qualitative approaches are needed within a holistic approach.

Many interventions' impact wanes when complete. Often those individuals that participated revert to previous maladaptive health behaviors. This can occur partly from a lack of a sense of ownership. Therefore, a holistic, structured approach is urgently needed, presented in a manner to enhance individual efficacy that enhances ownership. Strategies should also engage the expanded cancer survivor community thereby improving the health of the general cancer population, helping reduce existing cancer-related health disparities, and eliminating unnecessary costs on an already seriously strained public health system.

Here the investigators propose a 16-week pilot project to prove the feasibility and initial efficacy of such a holistic approach to optimize outcomes for the physical, mental and spiritual aspects of QOL as measured with standard instrumentation and qualitative self-report for 30 adult cancer survivors in the San Antonio, Texas area. The investigators will conduct pre, post and a six-month follow-up assessment for QOL.

DETAILED DESCRIPTION:
Here the investigators propose a pilot project to prove the concept and effectiveness of a holistic approach to optimize outcomes for physical, mental and spiritual aspects of QOL as measured with standard instrumentation and with qualitative self-report for 30 cancer survivors in the greater San Antonio, Texas area. The study team will achieve this urgently needed intervention by realization of the following three specific aims:

Specific Aim #1. Successfully engaging n=30 cancer survivors to complete a 16-week pilot intervention. The intervention will include a yoga-based regimen including meditation, an aerobic exercise program, diet improvement guidance coupled with psycho-social support text messaging based in Social Cognitive Theory to increase efficacy to promote health enhancing behaviors. For physical, mental and spiritual functioning outcome variables the study team will run a dependent -sample 't' test. For mental, spiritual outcome variables, single-systems analyses, will also be used to assess overall impact for each individual survivor as well as for the overall group as calculated in effect size. In addition, qualitative analyses from the survivor's self-reported perceptions of their levels of QOL will be analyzed using theme recognition. Investigators hypothesize that physical functioning will improve significantly (p< 0.05) and for the mental and spiritual primary outcome variables will result in at least a medium effect (d> 0.5) for the 30 cancer survivors when aggregated as a group.

Specific Aim #2. Demonstrating the feasibility that such an intervention can be implemented safely and cost-effectively for the cancer survivorship community. The study team will assess feasibility, by monitoring/recording all unexpected outcomes, adverse events, protocol deviations and compliance. Based on previous exercises studies the study team have completed, they hypothesize at least 90% compliance to the program coupled with no adverse events and will use these benchmarks by which to assess feasibility for the pilot.

Moreover, the study team will also record the total cost to deliver the intervention for the program and relate the cost back to benefit derived with metrics calculations for specific gains in physical, mental, and spiritual outcomes as well as an aggregate metric for overall QOL. Because the study team will be tabulating total cost, beyond just funded dollars, there is no set benchmark for feasibility but just offer the information as a metric for understanding true cost for a holistic approach.

Specific Aim #3. Monitoring the long-term impact for the survivors that complete the pilot for one six months after the 16-week intervention. The study team hypothesize that long term QOL outcomes will not change significantly as determined both by analyses of variance for physical functioning and single system analyses for the mental and spiritual measures from the time they complete the 16 weeks. Based on previous behavioral studies completed, the study team expect no more than 10% attrition to follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Have been given a diagnosis of any cancer in their lifetime; (active treatment or post treatment; but must be post diagnosis). (Even though the participant may be currently under treatment and limited in functionality, they will be included in the study as this pilot intervention is specifically intended to include any level of functionality, using a an individually designed program for optimizing outcome.)
* Have access or use of a mobile phone or computer to complete surveys and respond to text messages.
* Be able to speak understand English or Spanish.
* Oriented to time and place.

Exclusion Criteria:

* Currently enrolled in a competing protocol.
* Participants will be excluded it they present with any absolute contraindication to exercise testing as detailed by the American College of Sports Medicine Guidelines on Exercise Testing and Exercise Prescription 52. Specifically:
* Known significant change in the resting ECG suggesting significant ischemia.
* Recent myocardial infarction (within 2 days).
* Unstable angina.
* Uncontrolled cardiac arrhythmias causing symptoms or hemodynamic compromise.
* Severe symptomatic aortic stenosis.
* Uncontrolled symptomatic heart failure.
* Acute pulmonary embolus or pulmonary infarction.
* Acute myocarditis or pericarditis .
* Suspected or known dissecting aneurysm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-09-12 (Actual); Study Completion 2020-09-12 (Actual)

PRIMARY OUTCOMES:
Co-Morbidity Index | Weeks "0" and "16"
  Number of comorbidities
Motivational Style Profile | Weeks "0" and "16"
  The Apter Motivational Style Profile (AMSP) measures the dominance of all five pairs of metamotivational states identified in the theory: Telic vs. Paratelic, Autic vs. Alloic, Mastery vs. Sympathy, Negativism vs. Hedonism, and Locus of Control (Internal vs. External).
  The results of the AMSP questionnaire provide scores for different motivational dimensions, each representing a continuum between two opposing states. These scores indicate where an individual tends to fall on each continuum, reflecting their predominant motivational style.
  Each dimension has a pair of opposite states, and the scores on the AMSP indicate an individual's tendency toward one pole or the other of each pair. The higher the score on one pole, the more the person is inclined toward that style. Conversely, lower scores on the opposite pole indicate less preference for that state.
Quality of life (Medical Outcomes Short Form-36 (SF-36)) | Weeks "0" and "16"
  The SF-36 is often used as a measure of a person or population's quality of life. It comprises 36 questions that cover eight domains of health:
  1. Limitations in physical activities because of health problems
  2. Limitations in social activities because of physical or emotional problems
  3. Limitations in usual role activities because of physical health problems
  4. Bodily pain
  5. General mental health (psychological distress and well-being)
  6. Limitations in usual role activities because of emotional problems
  7. Vitality (energy and fatigue)
  8. General health perceptions
  Each of the eight domains has its own set of questions, with responses typically scored on a 0-100 scale (higher scores indicate better health). The scoring for each domain is as follows:
  0 represents the worst possible score (e.g., extreme limitation or poor health).
  100 represents the best possible score (e.g., no limitations or excellent health).
  After scoring each domain, two summary scores are calculated to prov
Level of pain | Weeks "0" and "16"
  The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be')
Non-Exercise Fitness Test | Weeks "0" and "16"
  The Jurca Non-Exercise Test is a simple and safe test to determine fitness level without having to do any exercise, using a regression equation using age, gender, body mass index (BMI), and self-reported physical activity levels to estimate VO2 max.
  VO2 Max is the maximum amount of oxygen the body can utilize during intense exercise, and it is considered one of the best indicators of aerobic fitness. The higher your VO2 max, the better your cardiovascular fitness.
Sleep Quality | Weeks "0" and "16"
  The Pittsburg Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. The PSQI consists of 19 individual items that are grouped into 7 components: Subjective Sleep Quality, Sleep Latency (Time Taken to Fall Asleep), Sleep Duration, Sleep Efficiency, Sleep Disturbances, Use of Sleep Medications, and Daytime Dysfunction.
  Each component assesses a specific aspect of sleep quality scored on a 0 to 3 scale based on the responses (higher scores indicating worse sleep quality). The total score for each component is calculated by adding the individual responses within that component. The scores are then summed to generate the PSQI global score, which helps classify sleep quality as "Good sleep quality" (0-4), "mild sleep problems" (5-10), "moderate sleep problems" (11-15), or "severe sleep problems" (16-21).
Perceived Stress | Weeks "0" and "16"
  The Perceived Stress Scale (PSS) is a measure of the degree to which situations in one's life are appraised as stressful. It focuses on how often a person feels overwhelmed, unable to cope, or unsure about their ability to handle challenges in the past month. It includes both the frequency and severity of perceived stressors.
  The PSS consists of 10 questions designed to assess feelings of unpredictability, lack of control, and feeling overwhelmed, as well as how often the individual felt nervous, upset, or helpless. Each item on the PSS is scored on a 5-point scale, ranging from 0 to 4: Never (0), Almost never (1), Sometimes (2), Fairly often (3), and Very often (4).
  The total score on the PSS indicates the level of perceived stress over the past month. Generally, the higher the score, the higher the perceived stress. PSS Score Ranges: 0-13: Low perceived stress, 14-26: Moderate perceived stress, and 27-40: High perceived stress.
Spiritual Well-being | Weeks "0" and "16"
  The Functional Assessment of Chronic Illness Therapy-Spiritual Well-being (FACIT-SP) consists of 12 items that assess two key dimensions of spiritual well-being:
  * Spiritual Well-Being: This measures the individual's sense of meaning and peace, connection to a higher power or a greater purpose, and the extent to which their spiritual beliefs contribute to their coping strategies and overall well-being.
  * Faith: This dimension measures how the individual's religious or spiritual beliefs help them make sense of their experiences and provide strength or comfort in times of adversity.
  Each of the 12 items is rated on a 5-point Likert scale, ranging from 0 to 4:
  0: Not at all (never true), 1: A little bit (rarely true), 2: Somewhat (sometimes true), 3: Quite a bit (often true), and 4: Very much (always true).
  Scores are summed to give a total spiritual well-being score. The total score typically ranges from 0 to 48, with higher scores indicating better spiritual well-being.
Exercise Barriers | Weeks "0" and "16"
  The Exercise Barriers Self-Efficacy (BSE) scores range from 0 to 100 for each item, with total or average scores calculated across multiple items.
  Interpretation:
  * Higher scores indicate greater confidence in overcoming barriers to exercising, such as time constraints or lack of motivation.
  * Lower scores suggest lower self-efficacy in handling challenges to exercise adherence.
Modeling of Exercise | Weeks "0" and "16"
  The Modeling of Exercise scores range varies, but often rated on a scale (e.g., 1 to 5 or 0 to 10) across several items related to observing others (e.g., family or friends) engaging in exercise. Total scores are summed or averaged.
  Interpretation:
  * Higher scores reflect greater exposure to role models for exercise, which could include parents, peers, or significant others.
  * Lower scores indicate less exposure to individuals modeling exercise behavior.
Exercise Self-Efficacy | Weeks "0" and "16"
  The Exercise Self-Efficacy (ESE) scores range from 0 to 100 for each item, with total or average scores calculated across multiple items.
  Interpretation:
  Higher scores denote greater confidence in one's ability to engage in regular exercise under various circumstances, such as bad weather or after a long workday.
  Lower scores imply a lack of confidence in maintaining exercise habits consistently.
Family support for exercise | Weeks "0" and "16"
  The Exercise Social Support Family (SSFA) scores are scaled responses from each item (e.g., 1 to 5 or 0 to 10), which are summed or averaged to create a total score.
  Interpretation:
  * Higher scores indicate greater perceived support from family members for exercise, such as encouragement, assistance, or participation.
  * Lower scores suggest limited family support for exercise behaviors.
Social support for exercise from peers | Weeks "0" and "16"
  The Exercise Social Support Friends (SSFR) scores are similar to SSFA: Scaled responses for each item (e.g., 1 to 5 or 0 to 10), summed or averaged to create a total score.
  Interpretation:
  * Higher scores reflect greater support from friends, such as exercising together or offering encouragement.
  * Lower scores indicate less perceived social support for exercise from peers.
Self-Identification as an Exerciser | Weeks "0" and "16"
  Likert scale scores (e.g., 1 to 7 or 1 to 10), summed or averaged to create a total score.
  Interpretation:
  * Higher scores represent stronger identification with being an exerciser, suggesting that exercise is a significant part of the individual's self-concept.
  * Lower scores indicate weaker identification with the identity of being an exerciser.
Body Image Scale | Weeks "0" and "16"
  The Body Image Scale for Cancer Survivors (BIS-C) asks patients to rate their body image on a scale of 0-3, with 0 meaning "not at all" (indicating no issue with body image), and 3 meaning "very much" (indicating significant body image concerns). The 10 items cover a range of topics, such as how satisfied the patient is with their appearance, how they feel about their body, and whether they find it difficult to look at themselves naked.
  Summary of BIS-C Score Ranges:
  0-10: Minimal body image concerns 11-20: Moderate body image concerns 21-30: Significant body image distress 31-40: Severe body image distress
Hope Scale | Weeks "0" and "16"
  The Adult Dispositional Hope Scale (ADHS) consists of 12 items and uses a Likert-type scale, with each item being rated from 1 ("Definitely False") to 8 ("Definitely True"). The items are divided into Agency and Pathways subscales, and the total score can be calculated by summing all items.
  Each item is rated on an 8-point scale, from 1 to 8, with 4 items measuring Agency and 4 items measuring Pathways. Some items are reverse-scored (e.g., negatively worded items). The possible range of scores for the ADHS is 12 to 96. Agency and Pathways scores range from 4 to 32.
  Interpretation of total scores: Low Hope (12 to 35), Moderate Hope (36 to 60), and High Hope (61 to 96).
  Subscale Interpretation: Higher Agency scores reflect stronger feelings of personal motivation and self-efficacy to initiate and sustain goal-directed actions; and higher score on the Pathways subscale reflects the belief that solutions and strategies are available to overcome obstacles and achieve goals.
Personal Meaningful Profile | Weeks "0" and "16"
  The Brief Personal Meaningful Profile (PMP-B) is intended to identify what really matters in the patient's life. It measures people's perception of personal meaning in their lives.
  The scale typically uses a Likert-type scale, often ranging from 1 to 5, where participants indicate how much they agree or disagree with statements about the meaningfulness of various aspects of their life (e.g., relationships, work, personal growth, etc.).
  Interpretation of Scores: Low Meaning (Lower Scores; 5-10), Moderate Meaning (Mid-Range Scores; 11-20), High Meaning (Higher Scores; 21-25)
Psychological distress and symptoms Inventory | Weeks "0" and "16"
  The Brief Symptom Inventory-18 (BSI-18) is a self-report checklist that measures psychological distress and symptoms. It contains 18 items across 3 key symptom domains (Somatization, Depression, Anxiety; 6 items in each), and is used to evaluate emotional functioning and identify the severity of psychological symptoms over a specified time period. Each item is rated on a 5-point Likert scale, reflecting the severity of symptoms over the past week.
  Minimum score: 0 (if the individual selects "Not at all" for every item). Maximum score: 72 (if the individual selects "Extremely" for every item).
  The BSI-18 is scored by summing the responses to all 18 items, with higher scores indicating significant distress. A score above 63 on any dimension is considered clinically significant.
Depression Scale | Weeks "0" and "16"
  The Center for Epidemiological Studies-Depression Scale (CES-D) is a 20-item measure that asks caregivers to rate how often over the past week they experienced symptoms associated with depression, such as restless sleep, poor appetite, and feeling lonely. Response options range from 0 to 3 for each item (0 = Rarely or None of the Time, 1 = Some or Little of the Time, 2 = Moderately or Much of the time, 3 = Most or Almost All the Time). Scores range from 0 to 60, with high scores indicating greater depressive symptoms.
Six-minute walk test (6MWT) | Weeks "0" and "16"
  The 6MWT is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
  The longer the distance covered, the better.
Balance | Weeks "0" and "16"
  Balance will be assessed while standing on a pressure mat with feet together, eyes opened and closed, for 30 seconds in each condition. Investigators will record data on the 'sway path distance' (displacement of the center of gravity in centimeters) in the two conditions. Longer distances indicate higher balance deficits.
Muscle strength | Weeks "0" and "16"
  * elbow flexors and shoulder elevators (i.e., upright row) isometric strength (in kilograms) will be tested using a strength dynamometer system in standardized positions;
  * Dominant hand grip strength in kilograms will be tested using a hand dynamometer;
  * Tests are performed three times and the best result is recorded.
Sit and reach test | Weeks "0" and "16"
  This test will be used to assess trunk and lower extremity flexibility. Test is performed three times and the best length is recorded.
Plasma concentration of inflammatory markers | Weeks "0" and "16"
  Baseline and end-of-study blood samples will be collected into K2-EDTA tubes and centrifuged to separate and aliquot plasma for subsequent cytokine protein analysis. Samples will be analyzed in duplicate using the Flex-Map 3D platform system (Luminex, Austin, TX) with the MILLIPLEX MAP Human Cytokine Panel A (HCYTA-60 K-08 with TNF-α, IL-1ra, IL-1β, IL-4, IL-6, IL-8, IL-10, and IFN-γ), Human Soluble Cytokine Receptor Panel (HSCRMAG-32 K-03 with sTNFRII, sTNFRII, and sIL-6R) and Milliplex-Human CVD Panel 3 with CRP (HCVD3MAG-67 K-01).
Real-time physical activity | Weeks "0" and "16"
  Physical activity will be measured by accelerometers (Actigraph GTX9, Actigraph, Inc. FL). Participants will be given the accelerometer one week prior to beginning the intervention to get their baseline physical activity levels. After the physical functional assessments, they will be given the accelerometers to wear on their wrist during the intervention to measure their changes in physical activity.

OTHER OUTCOMES:
Demographics | Weeks "0" and "16"
  Investigators will collect information on birthday, gender, ethnicity, race, highest level of education, current employment status, religion, marital status, how many children and their ages, and previous participation in yoga classes.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Health Promotion Research, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie the results reported in publications (including text, tables, figures, and appendices) will be shared with other researchers at UT Health San Antonio, with the NIH and on ClinicalTrials.gov
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available after summary result publication on ClinicalTrials.gov and when published in a peer review journal

REFERENCES:
- [Derived] Miller MJ, Hughes DC, Darby NT, Calderon T, Patel DI, Serra MC, Ramirez AG, Ortiz A, Almeida GJ. Balance Changes in Adult Cancer Survivors Participating in a 16-Week Therapeutic Yoga Program. Integr Cancer Ther. 2025 Jan-Dec;24:15347354241313048. doi: 10.1177/15347354241313048. PMID 39811878